CLINICAL TRIAL: NCT01934816
Title: Effects of KATP Channel Blockers on GLP-1 and Its Analogues' Mediated Microvascular Function
Brief Title: Incretin and KATP Channels
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical Issues with intervention
Sponsor: Katarina Kos (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor-Investigator, Katarina Kos, Senior Lecturer, Royal Devon and Exeter NHS Foundation Trust
Organization: Royal Devon and Exeter NHS Foundation Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2Myo2013; 1308823 (Registry Identifier: Trust Research and Development); 13/SW/0010 (Other: REC)
Record Dates: First submitted 2013-08-19; First posted 2013-09-04 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Healthy Subjects
Keywords: Incretins, KATP channels, intradermal injection
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glimepiride (Experimental): 4mg of Glimepiride once only before vascular testing and intradermal injections of GLP-1 and its analogues
  Interventions: Other: Intradermal injections of GLP-1 and its analogues
- Placebo tablet (Placebo Comparator): Placebo tablet is given in the morning of the intradermal injections of GLP-1 and its analogues
  Interventions: Other: Intradermal injections of GLP-1 and its analogues
- Glyburide (Active Comparator): 10mg of Glyburide before study visit and intradermal injections of GLP-1 and its analogues
  Interventions: Other: Intradermal injections of GLP-1 and its analogues

INTERVENTIONS:
Other: Intradermal injections of GLP-1 and its analogues — native GLP-1,Exenatide (Byetta)and Liraglutide (Victoza) will be microinjected at the same visit in no particular order in all study arms
  Other Names: microinjection of GLP-1 (native GLP-1); and its analogues such as Exenatide(Byetta); and Liraglutide (Victoza)

SUMMARY:
This study aims to examine the involvement of KATP channels on the microvascular actions of the incretin GLP-1 and its analogues in healthy individuals and to determine whether the acute oral administration of different KATP channel blockers which are oral medications for Type 2 diabetes such as Glibenclamide and Glimepiride differentially modulate the microvascular responses in these individuals.

DETAILED DESCRIPTION:
In addition to the glucose lowering effect, incretin based therapies have also an effect on the vascular system. Previous animal work and initial human studies suggest that incretins may be cardioprotective and act as vasodilators through opening of KATP channels.

Initial evidence suggests that beneficial vascular effects of incretin modifying agents may be nullified by the co-current treatment of the sulfonylurea (SU) drug glibenclamide. The investigators hypothesis is that the GLP-1 and SUs may have conflicting effects on the KATP channels and thus vascular function.

Interestingly the vascular actions of GLP-1 were not modified by a different treatment SUs called glimepiride, thereby raising the possibility that SUs differentially modulating the vascular actions of GLP-1 though this remains controversial.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 25 kg/m2

Exclusion Criteria:

* current or past history of diabetes (HbA1C more or equal 45mmol/mol)
* history of postprandial hypoglycaemia and dumping syndrome
* established cardiovascular disease
* established cerebrovascular disease
* blood pressure ≥ 140/85 mmHg
* Raynaud's disease
* severe impairment of renalhepatic, thyroid or adrenocortical function
* current treatment with any anti-hypertensive treatment
* lipid lowering therapy or systemic steroids
* lactation, pregnancy
* established vascular disease
* bariatric surgery
* significant weight change within the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in skin blood flow to GLP-1 and its analogues | 6 weeks
  Skin blood flow will be assessed before and after microinjection of GLP-1 or its analogues and the injection site monitored and compared to sites injected with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Kos, FRCP, PhD, Principal Investigator — University of Exeter
Locations (1):
- Royal Devon and Exeter NHS Foundation Trust, Exeter, United Kingdom